CLINICAL TRIAL: NCT01193738
Title: a Single Blind Cross Over Trial to Compare Osteopathic Compression of Pterygopalatine Node to Placebo Compression in Obstructive Sleep Apnea Syndrome.
Brief Title: Osteopathy and Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valerie Attali (Other)
Responsible Party: Sponsor-Investigator, Valerie Attali, MD, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2009-A01373-54; ADOREP 2009-068 (Other: ADOREP)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: osteopathy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- active osteopathic compression (Active Comparator): osteopathic compression of Pterygopalatine node
  Interventions: Procedure: osteopathic compression of Pterygopalatine node
- placebo osteopathic compression (Placebo Comparator): placebo osteopathic compression
  Interventions: Procedure: osteopathic compression of Pterygopalatine node

INTERVENTIONS:
Procedure: osteopathic compression of Pterygopalatine node — osteopathic compression of Pterygopalatine node

SUMMARY:
The main objective is to evaluate an osteopathic compression of pterygopalatine node on sleep obstructive apnea syndrome (OSA).

DETAILED DESCRIPTION:
Osteopathic compression will be compared to a placebo manoeuvre. Efficacy will be assessed by measuring pharyngeal collapsibility

ELIGIBILITY:
Inclusion Criteria:

* Male or Female aged 18 years or more
* obstructive sleep apnea syndrome with apnea/hypopnea index > or = 15/hour
* Body mass Index <40kg/m2

Exclusion Criteria:

* pregnant or lactating women
* participating to another trial
* acute infectious disease of upper respiratory airway tract at inclusion
* facial neuralgia at inclusion
* patients not able to stop treatment for OSA within one week before each visit
* allergy to latex
* dental extraction within 15 days before inclusion
* pharyngeal surgery in the past
* incapable adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
pharyngeal critical pressure | 30 minutes after osteopathic compression
  The collapsibility of the upper airway will be evaluated by pharyngeal critical pressure,assessed by measuring the intraluminal pressure associated with the cessation of airflow

SECONDARY OUTCOMES:
pharyngeal critical pressure | 48 hours
  The collapsibility of the upper airway will be evaluated by pharyngeal critical pressure,assessed by measuring the intraluminal pressure associated with the cessation of airflow
symptoms | 48 hours
  OSA symptoms
adverse events | 48 hours
  clinical evaluation of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: valerie attali, MD, Principal Investigator — Federation des pathologies du sommeil
Locations (1):
- Pathologies Du Sommeil Pitie Salpetriere, Paris, France

REFERENCES:
- [Derived] Jacq O, Arnulf I, Similowski T, Attali V. Upper airway stabilization by osteopathic manipulation of the sphenopalatine ganglion versus sham manipulation in OSAS patients: a proof-of-concept, randomized, crossover, double-blind, controlled study. BMC Complement Altern Med. 2017 Dec 20;17(1):546. doi: 10.1186/s12906-017-2053-0. PMID 29262824